CLINICAL TRIAL: NCT02327871
Title: Targeted Temperature Management With Therapeutic Hypothermia Using Esophageal COOLing After Cardiac Arrest: THE COOL STUDY
Brief Title: Esophageal Temperature Management After Cardiac Arrest
Acronym: THE-COOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IST cardiology (Industry)
Collaborators: Advanced Cooling Therapy LLC, d/b/a Attune Medical (Industry); Erik Kulstad, MD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDRCB 2014: AO-1145-42
Record Dates: First submitted 2014-12-24; First posted 2014-12-30 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Cardiac Arrest
Keywords: Therapeutic hypothermia; patients; Safety, Efficacy
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Esophageal cooling (Experimental): Specific treatment: The placement of the ECD will follow standard recommendations as per Instructions for Use. The ECD will be connected to the Gaymar console (Meditherm III, Gamida, France). In our institution, TH is performed in all patients resuscitated from an OHCA except those presenting exclusion criteria. TH can be initiated as soon as possible by administration of cold saline at 4°C if necessary followed by application of the available cooling device (blankets, endovascular methods, etc) aiming a target temperature of 32-34°C for 24 hours as recommended. 8-11,13 For all enrolled patient, the ECD will hereby replace the other cooling device usually used in our ICU.
  Interventions: Device: Esophageal cooling device (and usual standard procedure)

INTERVENTIONS:
Device: Esophageal cooling device (and usual standard procedure) — Standard treatments for resuscitation after CA will follow local, national, and international guidelines. Core temperature is measured using urinary Foley catheters and/or arterial temperature monitoring if available. During TH, sedation and analgesia is performed in routine. Neuromuscular blockade is induced to favor cooling and prevent shivering if necessary. Circulatory function is monitored by arterial catheter if necessary and blood pressure is maintained as usually. Hypotension is treated with dobutamine catecholamines titrated according cardiac output monitored using echocardiogram, or PiCCO® systems. Fluid management is left at the discretion of the attending physician. Prognostication after CA uses serial clinical examinations, biomarkers, transcranial Doppler, Electro-Encephalo-Gram, cerebral CT-scan or MRI, and/or Somato-Sensory-Evoked-Potential.
  Other Names: ECD

SUMMARY:
To control patient's body temperature remains of major importance especially after cardiac arrest (CA). Therapeutic hypothermia (TH) targeted to 32-34°C is now recommended for most unconscious CA patients. However, available modalities for inducing TH have a number of technical (side effects), logistical (difficulties of placement), and financial (cost) barriers. The Esophageal Cooling Device (ECD) is a multi-chambered silicone heat exchanger placed in the esophagus providing highly efficient heat transfer to a patient. The ECD is a device that potentially improves the effectiveness of TH in minimizing the risks of existing methods (such as invasive cooling). Initial mathematical and animal studies have shown strong support for the efficacy and safety of the ECD. Placement of a naso-gastric probe is a systematic standard of care for all unconscious patients suffering from CA. The present study will replace the usual naso-gastric probe by the ECD that can be used for gastric suctioning as usually done in such patients.

The aim of this prospective, interventional study is to assess the feasibility and safety of the ECD in resuscitated CA-patients and treated with 32-34°C targeted TH. The primary outcome is the feasibility of inducing, maintaining, and rewarming patients from TH using the ECD (cooling rate, rewarming rate, and the percent of time within goal temperature during the goal-temperature maintenance period). Evaluation of adverse events (including cardiac arrhythmias, severe bradycardia, myocardial infarction/re-infarction, dysphagia, odynophagia, aspiration pneumonia, non-aspiration pneumonia, esophageal reflux and injury, and esophagitis) will be closely monitored during the whole period of the targeted temperature management (secondary endpoint).

DETAILED DESCRIPTION:
Background The ability to control a patient's body temperature under a wide variety of conditions is extremely important, and is of particular importance after CA. TH targeted to 32-34°C as a targeted temperature management (TTM) demonstrably improves outcomes in at least two clinical conditions: adults resuscitated from CA and neonates suffering from hypoxic ischemic encephalopathy.1-7 TH is recommended for CA patients by major organizations that provide resuscitation guidelines, including the American Heart Association, the European Resuscitation Council, and the International Liaison Committee on Resuscitation.8-10 This indication was confirmed by a non-expert jury who provided clinical recommendations for five professional and international critical care societies (the American Thoracic Society, the European Respiratory Society, the European Society of Intensive Care Medicine, the Society of Critical Care Medicine, and the Société de Réanimation de Langue Française): the jury strongly recommends TTM to a target of 32-34°C as the preferred treatment (vs. unstructured temperature management) of out-of-hospital adult CA victims with a first registered electrocardiography rhythm of ventricular fibrillation or pulseless ventricular tachycardia and still unconscious after restoration of spontaneous circulation.11 Additional evidence exists, albeit lower level, for use of TH for comatose survivors of CA initially associated with non-shockable rhythms.8-10 The debate regarding the optimal level of TTM has been recently evaluated in a large randomized controlled trial comparing 2 different levels of TTM performed during 28 hours.12 In this study similar results regarding neuroprotection and survival have been obtained using either a 36°C target or a 33°C target (i.e. "real" TH).13 Consequently these 2 different levels of TTM can be used as it have been recently recalled by experts in the field. These treatments should be started as soon as possible, especially within the first 4 hours after CA. However this delay could be prolonged until 6 to 10 hours after CA.8-11 To date, however, available modalities for inducing precise TTM and TH have a number of technical, logistical, and financial barriers, including difficulties in placement, risks of use (such as needle sticks, infections, blood clots, and skin damage), and high cost. The Esophageal Cooling Device (ECD) is a disposable device that potentially improves the effectiveness of 32-34°C targeted TH while minimizing the risks of other existing methods such as invasive methods.14 The ECD is a multichambered silicone heat exchanger that is placed in the esophagus to provide highly efficient heat transfer to a patient while simultaneously maintaining access to the stomach to allow gastric suctioning, decompression, and drainage, as usually performed in such patients hospitalized in ICUs. The esophagus is in close proximity to blood flow from the heart and great vessels, and the ECD is designed to take advantage of this heat exchange environment. The ECD's ability to decompress the stomach and avoid distention of the esophagus away from the device ensures good contact with the esophageal mucosa, and thus maximizes heat transfer from the patient. The ECD replaces the standard gastric tube which is placed in the target patient population as a routine standard of care, is made of standard medical-grade silicone, and is generally similar in size and shape to the gastric tubes currently used. Initial mathematical and animal studies have shown strong support for the efficacy and safety of the ECD.14-16

Study design: Prospective, interventional study evaluating the feasibility (efficacy) and safety of the ECD in patients resuscitated from CA and treated with TH.

Patient population: Patient population will consist of patients suffering resuscitated out-of-hospital or in-hospital CA with stable return of spontaneous circulation (ROSC) and hemodynamic conditions with an indication to TH implementation according to standard recommendations.

Data collection: All clinical and biological parameters will be recorded according to the Utstein-style recommendations for reporting resuscitation outcomes. Neurologic outcome will be assessed according to the Cerebral Performance Category (CPC) score. Initial temperatures will be measured via a tympanic and naso-pharyngeal temperature sensors in the prehospital field and the inhospital cath-lab respectively. Continuous temperature measurement (specifically during cooling, maintenance, and rewarming) will be measured by bladder temperature sensors, and arterial temperature monitoring (Picco®) if available. Time of ECD placement and potential side effects will be recorded.

Specific treatment: The placement of the ECD will follow standard recommendations as per Instructions for Use. The ECD will be connected to the Gaymar console (Meditherm III, Gamida, France). In our institution, TH is performed in all patients resuscitated from an OHCA except those presenting exclusion criteria. TH can be initiated as soon as possible by administration of cold saline at 4°C if necessary followed by application of the available cooling device (blankets, endovascular methods, etc) aiming a target temperature of 32-34°C for 24 hours as recommended. 8-11,13 For all enrolled patient, the ECD will hereby replace the other cooling device usually used in our ICU.

Other treatments: Standard treatments for resuscitation after CA will follow local, national, and international guidelines as previously described. Briefly, core temperature is usually measured using esophageal or urinary Foley catheters with thermistor probe (Tyco Healthcare, France) and/or arterial temperature monitoring (PiCCO, Pulsion Medical System, France) if available and/or necessary. During TH, sedation is performed with continuous infusion of midazolam or propofol and sufentanil. Neuromuscular blockade is induced using cisatracurium to favor cooling and prevent shivering if necessary. Circulatory function is monitored by radial or femoral arterial catheter if necessary and blood pressure is maintained at ≥90mmHg systolic and >65mmHg mean arterial pressure. Hypotension is treated with dobutamine and norepinephrine or epinephrine titrated to the targeted blood pressure according to the cardiac output monitored using echocardiogram, or PiCCO® systems according to the physician in charge. Fluid management is left at the discretion of the attending physician. Neuromonitoring and prognostication after CA uses serial clinical examinations, biomarkers (lactates, creatinine, NSE, S100B protein), transcranial Doppler, daily Electro-Encephalo-Gram, cerebral CT-scan or MRI, and Somato-Sensory-Evoked-Potential if necessary.

Statistical analysis:

Since this is a pilot study a sample size of 15 patients was calculated based on local feasibility considerations. This is a non comparative study. Thus the statistical analysis will be descriptive. For all quantitative parameters, mean, SD, median and quartiles will be calculated. For qualitative parameters, percentage and their two-sided 95% confidence intervals will be calculated. All analyses will be made in patients who received the ECD. In case of unsuccessful attempt to use the ECD, the patient will be listed.

Informed consent and ethical considerations: This study will be conducted according to the principles of the Declaration of Helsinki of the World Medical Association. The protocol have been submitted, modified and accepted by the local Ethics Committee of our local AP-HP institution (Institutional Review Board of Paris VI Hospital, Comité de Protection des Personnes de GHPS, Paris 12ème, approval CPP/79-14, ID RCB 2014-A01145-42, 10/28/2014).

Written informed consent will be obtained before inclusion from each patient's next of kin when present at patient's admission.. According to French law and our local Ethics Committee and because of the short delay to enroll patients, if no family member can be reached before inclusion despite systematic researches performed by the physician in charge of the patient as soon as patient's admission, a patient presenting inclusion criteria and no exclusion criteria can be included in emergency. In all cases, surviving patients without severe neurological sequels will give their written informed consent as soon as possible (i.e. when awake).

An approval regarding the use of the ECD from the French committee responsible for the devices used in human beings (Agence Nationale de Sécurité du Médicament et des produits de santé, N° DMDTP/DMTECH/KB/2014-A01145-42, 9/4/2014) and the CE mark (N° , the 03/24/2014) have been specifically obtained separately. Specific insurances are delivered by ACT society and its French representing company IST Cardiology (Chubb Insurance Company of Europe SE, 10/10/2014, protocol 2014-A01145-42).

This trial has also been declared to the French Informatics' Society (Commission Nationale Informatique et Liberté N°1593420).

References:

1. HACA. Mild therapeutic hypothermia to improve the neurologic outcome after cardiac arrest. N Engl J Med. 2002;346(8):549-556.
2. Bernard SA, Gray TW, Buist MD, Jones BM, Silvester W, Gutteridge G, et al. Treatment of comatose survivors of out-of-hospital cardiac arrest with induced hypothermia. N Engl J Med. Feb 21 2002;346(8):557-563.
3. Shankaran S, Laptook AR, Poole WK. Hypothermia for perinatal asphyxial encephalopathy. N Engl J Med. Mar 18 2010;362(11):1051-1052; author reply 1052.
4. Sinclair HL, Andrews PJ. Bench-to-bedside review: Hypothermia in traumatic brain injury. Crit Care. Feb 15 2010;14(1):204.
5. Froehler MT, Ovbiagele B. Therapeutic hypothermia for acute ischemic stroke. Expert Rev Cardiovasc Ther. Apr 2010;8(4):593-603.
6. Dietrich WD, Bramlett HM. The Evidence for Hypothermia as a Neuroprotectant in Traumatic Brain Injury. Neurotherapeutics: The Journal of the American Society for Experimental NeuroTherapeutics. 2010;7(1):43-50.
7. Kelly FE, Nolan JP. The effects of mild induced hypothermia on the myocardium: a systematic review. Anaesthesia. May 2010;65(5):505-515.
8. Peberdy MA, Callaway CW, Neumar RW, Geocadin RG, Zimmerman JL, Donnino M, et al. Part 9: post-cardiac arrest care: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. Nov 2 2010;122(18 Suppl 3):S768-786.
9. Nolan JP, Neumar RW, Adrie C, Aibiki M, Berg RA, Bottiger BW, et al. Post-cardiac arrest syndrome: Epidemiology, pathophysiology, treatment, and prognostication A Scientific Statement from the International Liaison Committee on Resuscitation; the American Heart Association Emergency Cardiovascular Care Committee; the Council on Cardiovascular Surgery and Anesthesia; the Council on Cardiopulmonary, Perioperative, and Critical Care; the Council on Clinical Cardiology; the Council on Stroke. Resuscitation. 2008;79(3):350-379.
10. Nolan JP, Morley PT, Hoek TL, Hickey RW. Therapeutic hypothermia after cardiac arrest. An advisory statement by the Advancement Life support Task Force of the International Liaison committee on Resuscitation. Resuscitation. 2003;57(3):231-235.
11. Nunnally ME, Jaeschke R, Bellingan GJ, Lacroix J, Mourvillier B, Rodriguez-Vega GM, et al. Targeted temperature management in critical care: A report and recommendations from five professional societies. Crit Care Med. Dec 23 2010.
12. Nielsen N, Wetterslev J, Cronberg T, et al. Targeted Temperature Management at 33 degrees C versus 36 degrees C after Cardiac Arrest. N Engl J Med. 2013;369:2197-2206.
13. ILCOR statement on Nielsen study published in the N Engl J Med. http://www.med.upenn.edu/resuscitation/documents/TTMILCOR.pdf
14. Kulstad E, Metzger AK, Courtney DM, Rees J, Shanley P, Matsuura T, et al. Induction, maintenance, and reversal of therapeutic hypothermia with an esophageal heat transfer device. Resuscitation. Jul 1 2013.
15. Kulstad EB, Courtney DM, Waller D. Induction of therapeutic hypothermia via the esophagus: a proof of concept study. World J Emerg Med. 2012;3(2):118-122.
16. Vaicys V, Eason A, Schieber JD, Kulstad EB. Therapeutic hypothermia induction via an esophageal route-a computer simulation. Am J Emerg Med. Jul 2012;30(6):932-935.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age over 18 years)
* Successfully resuscitated from an out-of-hospital CA
* With sustained ROSC (ROSC maintained for >20/minutes)
* Admitted in the ICU
* Comatose (not obeying to verbal command)
* And treated with TH targeted to 32-34°C

Exclusion Criteria:

* Patient < 18 y.o.
* Patients with known esophageal deformity, or evidence of esophageal trauma, or previous esophageal disease (for example, known esophageal varices, cirrhosis, history of esophagectomy, previous swallowing disorders or dysphagia, achalasia, known ingestion of acidic or caustic poisons within the prior 24 hours etc.).
* Patients with less than 40 kg of body mass.
* Female patients known to be pregnant.
* Terminal disease or "do not resuscitate order" that could lead to early-onset therapeutic withdrawal (<48 hours after collapse).
* Unstable ROSC (defined as impossibility to maintain ROSC with palpable pulse for >20/minutes), or unstable hemodynamic conditions (defined as intractable severe cardiogenic shock or ECLS requiring) that could lead to multi-organ failure and early-onset death (<48 hours after collapse).
* Accidental hypothermia or hypothermia <30°C at admission
* Prolonged delay between CA and ROSC (i.e. time to ROSC > 60min)
* Prolonged delay between ROSC and inclusion > 360min
* Conscious patient (obeying to verbal command before starting TH)
* Severe bleeding or diathesis or uncontrolled hemorrhage before inclusion
* Esophageal bleeding before ECD insertion
* Pre-existing severe conductive disorder requiring pacing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The percent of time over the study period within 1°C of goal temperature (33°C) . | Targeted temperature management phase (TH) within the first 48 hours after inclusion

SECONDARY OUTCOMES:
Percentage of patients for whom the ECD maintained goal temperature +/-1°C for 85% of the time during the maintenance 33°C phase . | Targeted temperature management phase (TH) within the first 48 hours after inclusion
Composite adverse events including the following: cardiac arrhythmias, severe bradycardia, myocardial infarction/re-infarction, dysphagia, odynophagia, aspiration pneumonia, non-aspiration pneumonia, reflux, esophageal injury, and esophagitis. | Until three months (follow-up) after inclusion
Global and neurologic outcome will be assessed using the Overall (OPC) and the Cerebral Performance Category (CPC) score with blinded evaluation of the mid- and long-term neurological outcome | up to follow-up at 3 months after inclusion
  assessment by a independent physician unaware of the esophageal cooling

CONTACTS AND LOCATIONS:
Locations (1):
- Lariboisère, Paris, France